CLINICAL TRIAL: NCT01926951
Title: A Feasibility Study: An Evaluation of Renal Denervation Using Externally Focused Therapeutic Ultrasound With External Targeting and Tracking on Patients With Refractory Hypertension
Brief Title: Renal Denervation Using Externally Focused Therapeutic Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kona Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KM13-001
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal Denervation (Experimental): Renal Denervation using the Kona Surround Sound Externally Focused Therapeutic Ultrasound therapy.
  Interventions: Device: Surround Sound Externally Focused Therapeutic Ultrasound

INTERVENTIONS:
Device: Surround Sound Externally Focused Therapeutic Ultrasound — Externally Focused Therapeutic Ultrasound using the Kona Surround Sound System

SUMMARY:
This study will evaluate the effects of renal denervation using externally focused therapeutic ultrasound with external targeting and tracking on patients with refractory hypertension.

DETAILED DESCRIPTION:
This study is a prospective, multi-center trial wherein each included subject will receive the experimental externally focused ultrasound renal denervation therapy. It will be conducted on a maximum of twenty patients who meet the eligibility criteria and have signed the informed consent form.

Safety is the primary endpoint of this study. Safety will be assessed by incidence and evaluation of any serious adverse effects associated with the investigational procedure through the 52-week evaluation. Clinical utility is a secondary endpoint of this study. Clinical utility will be evaluated by comparing pre and post therapy systolic and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Average systolic blood pressure at least 160 mmHg
* Refractory, stable hypertension despite being treated with at least three hypertensive drugs
* Two functioning kidneys, defined as eGFR >= 45 ml/min
* At least one renal artery on each side which is greater than 4 mm.

Exclusion Criteria:

* History of nephrectomy or hydronephrosis
* Renal stenosis > 50%
* Renal stent
* Ambulatory blood pressure monitoring 24 hour average systolic blood pressure <= 135 mmHg
* Kidney stones which are symptomatic and/or > 1 cm
* History of abdominal surgery within the past 6 months
* Heterogeneities in the kidneys (cysts or tumors)
* Residual pyelonephritis
* History of myocardial infarction, unstable angina pectoris, or cerebrovascular accident within the last 6 months
* Hemodynamically significant valvular heart disease
* Implantable cardioverter defibrillator, pacemaker, neurostimulator or other device incompatible with MRI
* Body weight > 150 kilograms
* Target treatment depth > 14 cm from the skin line
* Pregnant, nursing or intends to become pregnant during the trial period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety | 52-week post-treatment
  Safety will be assessed by incidence and evaluation of any serious adverse effects associated with the investigational procedure through 52-week evaluation. Included in this assessment will be the proportion of subjects with any of the following outcomes: 1) death, or 2) medical morbidity.

SECONDARY OUTCOMES:
Clinical Utility | 52-week post-treatment
  Clinical utility will be evaluated by comparing pre and post therapy systolic and diastolic blood pressure.

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (2):
  - St. Anne's University Hospital, Brno
  - Nemocnice Na Homolee Hospital, Prague
- Mercy Angiography, Aukland, New Zealand